CLINICAL TRIAL: NCT04861688
Title: A Randomized Double-blind, Placebo-controlled, Multi-center Trial to Investigate the Efficacy and Safety of NeuroAiD II™ (MLC901) to Improve Cognitive Functioning in Non-surgical Mild Traumatic Brain Injury Patients
Brief Title: NeuroAiD II™ (MLC901) in Mild Traumatic Brain Injury
Acronym: SAMURAI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Moleac Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFSA2020_03
Record Dates: First submitted 2021-04-19; First posted 2021-04-27 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Randomized Double-blind; Placebo-controlled; NeuroAiD II™; MLC901; Traditional Chinese Medicine; Cognitive Functioning
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Medicine, Chinese Traditional; Neuroaid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeuroAiD II™ (MLC901) (Active Comparator): Recommended treatment is 2 capsules orally, 3 times a day (i.e. 6 capsules per day). Treatment is 12 weeks.
  Interventions: Combination Product: Traditional Chinese Medicine (NeuroAiD II™ (MLC901)
- Placebo (Placebo Comparator): Capsule 2 capsules orally, 3 times a day
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Traditional Chinese Medicine (NeuroAiD II™ (MLC901) — NeuroAiD II™ (MLC901) contains the extracts of 9 botanical active ingredients blended with commonly used excipients. The 9 botanical active ingredients are traditional herbs well documented in the Pharmacopoeia of the People's Republic of China.
  Arms: NeuroAiD II™ (MLC901)
Other: Placebo — Placebo with same appearance as active intervention
  Arms: Placebo

SUMMARY:
A Randomized Double-blind, Placebo-controlled, Multi-center Trial to determine the efficacy of NeuroAiD II™ (MLC901) in improvement of cognitive functioning of adult patients with long-term cognitive impairment following mild traumatic brain injury (mTBI) and to assess safety of NeuroAiD™ (MLC901) in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with mild TBI, which occurred 1-12 months prior enrolment to the study. Mild TBI is defined as an external force from an incident causing injury to the brain and resulting in an altered level of consciousness. The mTBI diagnosis should be documented. Mild TBI is evidenced by any of the following:

   * best Glasgow Coma Score 13-15 as assessed on scene, on admission and over next 3 days
   * loss of consciousness for up to 30 minutes
   * dazed and confused at the time of injury or post-TBI amnesia of < 24 hours duration.
2. Patient experiencing cognitive impairment following injury, determined by the Cognitive Failures Questionnaire score >30.
3. Adult male or female patients aged 18-65 years.
4. The patient has signed an Informed Consent form (ICF) for participation in this study before initiation of study procedures.
5. The patient can understand all protocol requirements, perform the study procedures, and agree to all limitations specified in the protocol.
6. The patient agrees to use adequate contraception methods.

Exclusion Criteria:

1. Moderate or Severe TBI, determined by best Glasgow Coma Score of <13 (as assessed on scene, on admission and over next 3 days), or injury requiring neurosurgery (even if surgery was not done)
2. Co-existing severe co-morbidity, including end stage renal failure, spinal cord injury, significant substance abuse, severe liver disease, significant mental illnesses, diabetes requiring insulin injections, severe agitation, advanced cancer or other severe conditions with life expectancy of less than 5 years. The decision on significance of the comorbidity for inclusion/exclusion from current study is made by the Investigator.
3. Current participation in another clinical trial within 30 days.
4. Women who are pregnant or who have a positive urine pregnancy test or breast-feeding.
5. Not fluent in Russian language or have aphasia/dysphasia.
6. No documented evidence of mTBI.
7. Known allergy to MLC901/NeuroAiD II™ or any of its component ingredients.
8. Other medical condition which in the opinion of the Principal Investigator would place undue risk on the patient if included in the trial or likely to interfere with NeuroAiD II™.
9. History of psychic (including depressive) disorders, physical and other factors that do not allow for adequate self-assessment of one's behaviour and for compliance with the protocol requirements, including history of psychiatric disorders.
10. Use of hormonal contraceptives, either oral or implant*.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Central Nervous System Vital Signs (CNS-VS), Domain score: Complex Attention | 6 months of treatment compared to baseline
  Change in complex attention score, determined using Central Nervous System Vital Signs (CNS-VS) computer cognitive testing system, after 6 months of treatment compared to baseline in the group of patients receiving NeuroAiD II™ (MLC901), compared to the placebo group.
  In the domain dashboard, above average domain scores indicate a Standard Score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-102 or PR 25-74, indicating normal function. Low average is SS 80-99 or PR 9-24 indicating a slight deficit or impairment. Below average is SS 70-79 or PR 2-8, indicating moderate level of deficit or impairment. Very low is SS less than 70 or a PR less than 2, indicating a deficit and impairment. Lower score is better for Complex Attention.

SECONDARY OUTCOMES:
CNS-VS system, Domain score: Execution Function | after 6 months of treatment compared to baseline
  Changes in the scores for the following cognitive domains: executive functioning, determined by CNS-VS system, after 6 months of treatment compared to baseline, in the NeuroAiD II™ (MLC901) group, compared to the placebo group.
  In the domain dashboard, above average domain scores indicate a Standard Score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-102 or PR 25-74, indicating normal function. Low average is SS 80-99 or PR 9-24 indicating a slight deficit or impairment. Below average is SS 70-79 or PR 2-8, indicating moderate level of deficit or impairment. Very low is SS less than 70 or a PR less than 2, indicating a deficit and impairment. Higher score is better.
CNS-VS system, Domain score: Processing speed | after 6 months of treatment, compared to baseline
  Changes in the scores for the following cognitive domains: processing speed, determined by CNS-VS system, after 6 months of treatment compared to baseline, in the NeuroAiD II™ (MLC901) group, compared to the placebo group.
  In the domain dashboard, above average domain scores indicate a Standard Score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-102 or PR 25-74, indicating normal function. Low average is SS 80-99 or PR 9-24 indicating a slight deficit or impairment. Below average is SS 70-79 or PR 2-8, indicating moderate level of deficit or impairment. Very low is SS less than 70 or a PR less than 2, indicating a deficit and impairment. Higher score is better.
CNS-VS system, Domain score: Visual memory | after 6 months of treatment, compared to baseline
  Changes in the scores for the following cognitive domains: visual memory, determined by CNS-VS system, after 6 months of treatment compared to baseline, in the NeuroAiD II™ (MLC901) group, compared to the placebo group.
  In the domain dashboard, above average domain scores indicate a Standard Score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-102 or PR 25-74, indicating normal function. Low average is SS 80-99 or PR 9-24 indicating a slight deficit or impairment. Below average is SS 70-79 or PR 2-8, indicating moderate level of deficit or impairment. Very low is SS less than 70 or a PR less than 2, indicating a deficit and impairment. Higher score is better.
CNS-VS system, Domain score: Verbal memory | after 6 months of treatment, compared to baseline
  Changes in the scores for the following cognitive domains: verbal memory, determined by CNS-VS system, after 6 months of treatment compared to baseline, in the NeuroAiD II™ (MLC901) group, compared to the placebo group.
  In the domain dashboard, above average domain scores indicate a Standard Score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-102 or PR 25-74, indicating normal function. Low average is SS 80-99 or PR 9-24 indicating a slight deficit or impairment. Below average is SS 70-79 or PR 2-8, indicating moderate level of deficit or impairment. Very low is SS less than 70 or a PR less than 2, indicating a deficit and impairment. Higher score is better.
CNS-VS system, Domain score: Reaction time | after 6 months of treatment, compared to baseline
  Changes in the scores for the following cognitive domains: reaction time, determined by CNS-VS system, after 6 months of treatment compared to baseline, in the NeuroAiD II™ (MLC901) group, compared to the placebo group.
  In the domain dashboard, above average domain scores indicate a Standard Score (SS) greater than 109 or a Percentile Rank (PR) greater than 74, indicating a high functioning test subject. Average is a SS 90-102 or PR 25-74, indicating normal function. Low average is SS 80-99 or PR 9-24 indicating a slight deficit or impairment. Below average is SS 70-79 or PR 2-8, indicating moderate level of deficit or impairment. Very low is SS less than 70 or a PR less than 2, indicating a deficit and impairment.Lower score is better.
Rivermead Post Concussion Symptoms Questionnaire (RPQ) | after 6 months of treatment, compared to baseline
  Change in the Rivermead Post Concussion Symptoms Questionnaire (RPQ) total score, after 6 months of treatment, compared to baseline, in the NeuroAiD II™ (MLC901) group compared to the placebo group.
  Scoring system is in two groups. RPQ-3 is potentially 0-12 and a higher score is worse, requires closer monitoring. RPQ-13 score is potentially 0-52 where higher scores reflect greater severity.

CONTACTS AND LOCATIONS:
Locations (4):
- Russia (4):
  - Nizhny Novgorod regional clinical hospital named after N. A. Semashko, Nizhny Novgorod
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Municipal Polyclinic № 106 of St.Petersburg, Saint Petersburg
  - X7 Research, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pilipenko PI, Ivanova AA, Kotsiubinskaya YV, Grigoryeva VN, Khrulev AY, Skorokhodov AV, Gavrik MM, Mkrtchan NN, Majdan M, Valkovic P, Rabarova D, Barker-Collo S, Jones K, Feigin VL. A double-blind, placebo-controlled, randomized, multi-centre, phase III study of MLC901 (NeuroAiDTMII) for the treatment of cognitive impairment after mild traumatic brain injury. PLoS One. 2025 Jul 10;20(7):e0310229. doi: 10.1371/journal.pone.0310229. eCollection 2025. PMID 40638707
- [Derived] Pilipenko P, Ivanova AA, Kotsiubinskaya YV, Feigin V, Majdan M, Grigoryeva VN, Khrulev AY. Randomised, double-blind, placebo-controlled study investigating Safety and efficAcy of MLC901 in post-traUmatic bRAin Injury: the SAMURAI study protocol. BMJ Open. 2022 Apr 13;12(4):e059167. doi: 10.1136/bmjopen-2021-059167. PMID 35418437